CLINICAL TRIAL: NCT07304453
Title: Combination Therapy With Nucleo CMP and Neurorubine Provides Sustained Long-term Pain Control Compared to Carbamazepine in Classical Trigeminal Neuralgia: A Randomized Clinical Trial
Brief Title: Nucleo CMP and Neurorubine Versus Carbamazepine for Classical Trigeminal Neuralgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karbala University (Other)
Responsible Party: Principal Investigator, Salah M. Ibrahim, Chief oral surgery department, Kufa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Classical Trigeminal Neuralgia
Record Dates: First submitted 2025-11-25; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Trigeminal Neuralgia; Neuropathic Pain
Keywords: Trigeminal Neuralgial; Nucleo CMP; Neurorubine; Carbamazepine
MeSH Terms: conditions — Trigeminal Neuralgia; Neuralgia

STUDY DESIGN:
Intervention Model Description: Allocation:
  Randomized
  Intervention Model:
  Parallel Assignment
  Masking:
  Single (Outcomes Assessor)
  Primary Purpose:
  Treatment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Carbamazepine Therapy (Active Comparator): Participants received conventional carbamazepine tablets administered orally with meals. Treatment was initiated at 100 mg twice daily, with dose titration based on clinical response and tolerability up to a maximum of 400 mg twice daily.
  Interventions: Drug: Conventional Carbamazepine Therapy
- Nucleo CMP and Neurorubine Combination (Experimental): participants received a combination regimen administered orally with meals. During Weeks 1-6, patients took two capsules of Nucleo CMP daily plus two tablets of Neurorubine daily. During Weeks 7-9 (maintenance phase), patients took one tablet of Neurorubine daily.
  Interventions: Drug: Nucleo CMP and Neurorubine Combination

INTERVENTIONS:
Drug: Conventional Carbamazepine Therapy — Carbamazepine (Control): An anticonvulsant that acts primarily by blocking sodium channels to reduce nerve hyperexcitability. It provides symptomatic relief by suppressing pain transmission.
  Arms: Conventional Carbamazepine Therapy
Drug: Nucleo CMP and Neurorubine Combination — Nucleo CMP + Neurorubine (Experimental): A combination of nucleotides (cytidine monophosphate) and neurotropic B-vitamins (B1, B6, B12). This intervention aims to be neuroregenerative, promoting myelin formation and axonal repair rather than just suppressing pain signals.
  Arms: Nucleo CMP and Neurorubine Combination

SUMMARY:
Trigeminal neuralgia is a severe facial pain condition that significantly impacts quality of life. While the standard medication, carbamazepine, provides relief, it is often associated with side effects and rapid pain recurrence upon discontinuation. This randomized clinical trial compares the efficacy and safety of conventional carbamazepine therapy against a novel combination therapy consisting of Nucleo CMP (cytidine monophosphate) and Neurorubine (Vitamin B complex). The study aims to evaluate pain reduction during active treatment and the sustainability of pain control after treatment cessation.

DETAILED DESCRIPTION:
Trigeminal neuralgia (TN) is a severe neuropathic pain disorder characterized by paroxysmal electric shock-like pain in the trigeminal nerve distribution. While anticonvulsants, particularly carbamazepine, are the first-line treatment, they often provide incomplete relief, are associated with dose-limiting side effects (sedation, dizziness), and may lead to tolerance over time. This study investigates a novel therapeutic approach targeting nerve regeneration rather than solely symptom suppression.

This randomized, assessor-blinded, parallel-group, active-controlled clinical trial evaluates the efficacy, safety, and long-term sustainability of a combination therapy consisting of Nucleo CMP (cytidine monophosphate) and Neurorubine (Vitamin B complex: B1, B6, B12) compared to conventional carbamazepine therapy.

The study enrolled 38 patients diagnosed with classical trigeminal neuralgia according to International Headache Society criteria. Participants were randomized to one of two arms:

Control Group: Received Carbamazepine initiated at 100mg twice daily, titrated based on response and tolerability up to 400mg twice daily.

Intervention Group: Received a combination protocol. For weeks 1-6, participants took two capsules of Nucleo CMP and two tablets of Neurorubine daily. For weeks 7-9, participants entered a maintenance phase taking one tablet of Neurorubine daily.

The primary objective is to assess pain reduction using the Visual Analogue Scale (VAS). Secondary objectives include the frequency of pain attacks per day, safety/tolerability profiles, and the sustainability of pain control following the cessation of active treatment. Assessments were conducted at baseline, 3 weeks, 6 weeks, and 3 weeks following treatment cessation. The study hypothesizes that the neuroprotective and neuroregenerative properties of the combination therapy will provide superior sustained pain control compared to the symptomatic relief provided by carbamazepine.

ELIGIBILITY:
Inclusion Criteria:

.• Age between 18-80 years

* Clinical diagnosis of classical trigeminal neuralgia according to International
* Headache Society (IHS) diagnostic criteria
* Pain duration of at least 3 months
* Baseline Visual Analogue Scale (VAS) pain score greater than or equal to 4
* Ability to provide informed consent and comply with study procedures
* No contraindications to study medications

Exclusion Criteria:

* Secondary trigeminal neuralgia due to underlying pathology
* Atypical facial pain or other orofacial pain conditions
* Significant cardiovascular, hepatic, or renal disease
* Pregnancy or lactation
* Current use of anticonvulsants or other neuropathic pain medications
* History of allergic reactions to study medications
* Cognitive impairment preventing reliable pain assessment
* Concurrent participation in other clinical trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-01-07 (Actual); Primary Completion 2024-07-14 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity Visual Analogue Scale (VAS) Score | Baseline, Week 3, Week 6, and Week 9 (3 weeks post-treatment cessation)
  Pain intensity was assessed using a standardized 10-point Visual Analogue Scale (VAS). Patients indicated their pain level on a continuous line anchored by 0 and 10, where 0 represents "no pain" and 10 represents "worst possible pain." Higher scores indicate greater pain intensity. Assessments were recorded at Baseline, Week 3, Week 6, and Week 9 (3 weeks post-treatment cessation).

SECONDARY OUTCOMES:
Frequency of Pain Attacks | Baseline, Week 3, Week 6, and Week 9 (3 weeks post-treatment cessation)
  The average number of paroxysmal pain attacks occurring per day, recorded by patients in daily diaries. Higher numbers indicate higher disease burden.

CONTACTS AND LOCATIONS:
Locations (1):
- Oral Medicine Clinic, College of Dentistry, University of Kerbala, Karbala, Kerbala, Iraq